CLINICAL TRIAL: NCT03376412
Title: A Prospective Study to Evaluate the Raindrop Near Vision Inlay in Presbyopes Implanted Under a Corneal Flap or Within a Small-Incision Pocket
Brief Title: A Study to Evaluate the Raindrop Near Vision Inlay Under Flap or Within Pocket
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Whitten Laser Eye (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDR2017-004
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: The study will be a prospective, single-center, open label clinical trial where a maximum of 60 consecutive non-dominant eyes are implanted with the Raindrop Near Vision Inlay.
Masking Description: No Masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm Treatment. (Experimental): All patients will be unilaterally implanted in the non-dominant eye with the Raindrop Near Vision Inlay for the compensation of presbyopia.
  Interventions: Device: Raindrop Near Vision Inlay

INTERVENTIONS:
Device: Raindrop Near Vision Inlay — A maximum of 60 consecutive non-dominant eyes will be implanted with the Raindrop Near Vision Inlay.

SUMMARY:
The objective of this study is to evaluate the Raindrop® Near Vision Inlay for the improvement of near vision in presbyopes implanted under a corneal flap or within a small-incision pocket.

DETAILED DESCRIPTION:
Patients must require a reading add from +1.5 to +2.5 D, and both emmetropes as well as ametropes (requiring concurrent LASIK) are included in the investigation. Suitable patients will undergo implantation of the Raindrop inlay in the non-dominant eye to improve near vision. If necessary, a LASIK excimer ablation will first be performed to optimize postoperative vision at near and distance. Patients will follow a one-month regimen of strong steroid, at a minimum, after corneal inlay implantation to facilitate healing and visual recovery.

ELIGIBILITY:
Inclusion Criteria:

1.1.1 Patients require a near reading add from +1.5 to +2.5 D in the non-dominant eye.

1.1.2 Patients have a photopic pupil size of at least 3.0 mm in the non-dominant eye.

1.1.3 Patients have a central corneal thickness ≥ 500 microns in the non-dominant eye.

1.1.4 Patients have corrected distance and near visual acuity of 20/25 or better in each eye.

1.1.5 Patients have uncorrected near acuity of 20/40 or worse in the non-dominant eye.

1.1.6 Patients are willing and able to understand and sign a written Informed Consent Form prior to any study-specific procedures.

1.1.7 Patients are willing and able to return for scheduled follow-up examinations for 24 months after corneal inlay implantation.

Exclusion Criteria:

1.1.1 Patients with clinically significant dry eye (i.e., significant diffuse punctate staining with fluorescein and a tear breakup time less than 8 s) in either eye.

1.1.2 Patients with a planned corneal residual bed thickness that is less than 250 microns (corneal thickness - (intended flap thickness + intended ablation depth)).

1.1.3 Patients with macular pathology based on dilated fundus exam and/or optical coherence tomography (OCT) image.

1.1.4 Patients who would be co-managed by an ophthalmologist or optometrist who is not approved as a ReVision Optics investigator.

1.1.5 Patients with ocular pathology or disease (including pupil pathology such as fixed pupils) that might confound the outcome or increase the risk of adverse event.

1.1.6 Patients taking systemic or topical medications that might confound the outcome or increase the risk of adverse event. Patients taking isotretinoin or amiodarone hydrochloride and any other medication that affects the tear film or accommodation, including but not limited to, mydriatic, cycloplegic and mitotic agents, tricyclic, phenothiazines, benzodiazepines, and first generation antihistamines.

1.1.7 Patients with known sensitivity to any planned study medications. 1.1.8 Patients with residual, recurrent, active or uncontrolled eyelid disease. 1.1.9 Patients with significant corneal asymmetry or irregular topography. 1.1.10 Patients with clinically significant anterior segment pathology. 1.1.11 Patients with any corneal abnormality, including but not limited to, slit lamp findings for corneal staining Grade 3 or higher, recurrent corneal erosion or severe basement membrane disease, and pterygium extending onto the cornea.

1.1.12 Patients with ophthalmoscopic/topographic signs of keratoconus or those who are keratoconus suspect.

1.1.13 Patients with history of Herpes zoster or Herpes simplex keratitis. 1.1.14 Patients with any progressive retinal disease or patients with a history or evidence of retinal vascular occlusion and/or hypercoagulability, because of the risks associated with high pressures during suction application.

1.1.15 Patients with known history of steroid-responsive intraocular pressure increases, glaucoma, preoperative IOP > 21 mm Hg, or are otherwise suspected of having glaucoma.

1.1.16 Patients with amblyopia or strabismus or those who are at risk for developing strabismus postoperatively as determined by corneal light reflex and cover-uncover testing.

1.1.17 Patients with diabetic retinopathy, collagen, vascular, diagnosed autoimmune disease (e.g., lupus, rheumatoid arthritis, fibromylagia), immunodeficiency (e.g., HIV), connective tissue disease, or clinically significant atopic syndrome such as allergies or asthma.

1.1.18 Patients on chronic systemic corticosteroid or other immunosuppressive therapy that may affect wound healing.

1.1.19 Patients with any type of active cancer (ophthalmic or non-ophthalmic). 1.1.20 Patients with uncontrolled infections of any kind. 1.1.21 Patients who are pregnant, lactating, of child-bearing potential and not practicing a medically approved method of birth control, or planning to become pregnant during the course of the trial, and patients with other conditions associated with fluctuation of hormones that could lead to refractive changes.

1.1.22 Patients who actively participate in contact sports (i.e., boxing, martial arts) where impacts to the face and eye are a normal occurrence.

1.1.23 Patients participating in any other ophthalmic or non-ophthalmic drug/device clinical trials during the time of this clinical investigation.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-08 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Visual Acuity | 24 Months
  After the inlay procedure, patients will attain functional near acuity in the inlay eye and functional distance vision binocularly.

SECONDARY OUTCOMES:
Incidence of Corneal Reaction | 24 Months
  Patients implanted either under a corneal flap or within a small-incision pocket will have minimal incidence of corneal reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mark E. Whitten, MD, Principal Investigator — Whitten Laser Eye
Locations (1):
- Whitten Laser Eye, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No